CLINICAL TRIAL: NCT05468645
Title: In Vivo Mass Balance Study of a Single Oral Dose of [14C]Hemay005 in Healthy Chinese Male Adults
Brief Title: In Vivo Mass Balance Study of [14C]Hemay005
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ganzhou Hemay Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HM005MB1S01/CRC-C2209
Record Dates: First submitted 2022-06-15; First posted 2022-07-21 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Health Volunteer

STUDY DESIGN:
Intervention Model Description: The subjects fast for at least 10 h before dosing, take orally a suspension prepared with 60 mg of [14C]Hemay005 (approximately 100 µCi of radioactivity) and 240 mL of water, and then fast for another 4 h after dosing. One hour of water deprivation is required respectively before and after dosing (except water for dosing).
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C]Hemay005 (Experimental)
  Interventions: Drug: [14C]Hemay005

INTERVENTIONS:
Drug: [14C]Hemay005 — Name: [14C]Hemay005 Dose: 60 mg/100 µCi Storage: store at -10℃ to -30 °C, tightly closed and protected from light.

SUMMARY:
This study is a single-center, single-dose, non-randomized, open-label study to evaluate the in vivo mass balance of [14C]Hemay005. Six healthy male subjects are planned to be enrolled.

DETAILED DESCRIPTION:
The subjects are examined during the screening period (D-14 to D-2) and those who are qualified for the preliminary assessment are admitted to the clinical research center after qualification against the inclusion and exclusion criteria (D-2). After admission, they are trained on medication, urine and feces collection and other procedures to make sure that they can perform relevant operations according to the requirements of the protocol and corresponding operation manuals or procedures. Random urine and feces specimens (-24 h-0 h) are collected before dosing (D-1) and the subjects are deprived of food for at least 10 h and water for 1 h before dosing. On the morning of the first day of the study (D1), blood specimens are collected within 1 h before dosing, and the investigational product is taken orally on an empty stomach. The subjects are deprived of food for 4 h and water for 1 h after dosing. All urine and feces specimens excreted within the specified time intervals of 0-240 h and blood specimens sampled at specified time points within 0-168 h after dosing are collected. Phased testing is adopted in this study to determine whether specimen collection may be terminated in advance or the collection time needs to be prolonged based on the test results. If the specimen collection time exceeds that tentatively specified in the protocol, the collection should be extended at an interval of 24 h (urine, feces) or an integer multiple interval of 24 h (blood specimen) until the criteria for termination of specimen collection specified in the protocol are met. Meanwhile, the safety monitoring is continued until the completion date of the specimen collection.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand the objectives and requirements of this study; willing to participate in the clinical study and sign the informed consent form; capable of communicating with investigators and completing the entire study as required;
2. Healthy male subjects between the ages of 18-40 years (inclusive), with normal defecation (1-2 times a day);
3. Body weight ≥ 50 kg, BMI: 19.0-26.0 kg/m2 (inclusive);
4. Normal or abnormal but clinically insignificant results of vital signs, physical examination, laboratory tests (routine hematology, blood biochemistry, coagulation function, routine urinalysis, thyroid function, routine stool test + occult blood, etc.), 12-lead ECG, chest X-ray (posterior-anterior), and abdominal B-mode ultrasound (liver, gallbladder, pancreas, spleen, kidney, bladder);
5. Male subjects of reproductive potential who promise to maintain no fathering or sperm donation plan, and voluntarily take effective contraceptive measures (such as complete abstinence, condom, contraceptive sponge, contraceptive gel, contraceptive film, intra-uterine contraceptive device, oral or injectable contraceptive, subcutaneous contraceptive implant, etc.) (contraceptive methods are detailed in Appendix 3) from admission to 6 months after the last dose.

Exclusion Criteria:

1. Allergic constitution or allergic diseases, or known allergies to the ingredients, similar products or excipients of the investigational product;
2. Hemorrhoids or perianal diseases with regular/ongoing hematochezia, habitual constipation or diarrhea, irritable bowel syndrome (IBS), inflammatory bowel disease and other diseases that affect the absorption, distribution, metabolism and excretion of oral drugs, or the safety evaluation of the investigational product; history of severe vomiting and diarrhea within 7 d before dosing;
3. Previous history of peptic ulcer or bleeding, or any serious disease or condition that may affect the study results in the opinion of the investigators, including but not limited to disorders of the skin and mucous membrane, eyes, ears, noses, throat, circulatory system, endocrine system, respiratory system, nervous system, digestive system, urinary system, blood, immune, mentality, or metabolism, or chronic infectious diseases (such as tuberculosis).
4. Positive for hepatitis B surface antigen, hepatitis C antibody, human immunodeficiency virus, or treponema pallidum antibody;
5. Reception of major surgery within 6 months before dosing, or scheduled for a surgery during the study;
6. History of drug abuse, or use of dope within 3 months before dosing, or positive for urine drug abuse screening;
7. Mean smoking quantity > 10 cigarettes/d 3 months before dosing;
8. Regular drinkers within 3 months before dosing, that is, drinking volume > 14 U of alcohol per week (1 U = 360 mL beer or 45 mL spirits with 40% alcohol or 150 mL wine); positive breath alcohol test result;
9. Blood loss or blood donation ≥ 400 mL within 3 months before dosing, or blood transfusion within 1 month before dosing;
10. Use of any drug that inhibits or induces liver drug metabolism enzymes within 1 d before dosing (see Appendix 1 for details);
11. Use of any prescription drugs, over-the-counter drugs, Chinese herbal medicines or food supplements, such as vitamins and calcium supplements, within 14 d before dosing; participation in clinical trials of other drugs and reception of the investigational product within 3 months before dosing;
12. Vaccination within 1 month before dosing or scheduled for a vaccination during the study;
13. Special dietary requirements or unable to follow a uniform diet; history of needle or blood sickness, difficulty in blood collection, or intolerance of venipuncture blood collection;
14. Long-term exposure to radioactivity, significant radioactive exposure (≥ 2 chest/abdomen CTs, or ≥ 3 other types of X-ray examinations); participation in radiolabeled drug trials within 1 year before dosing;
15. ther factors that render the subjects unsuitable for participating in this study (determined by the investigators).

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2022-07-25 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
pharmacokinetic (PK) profile of Hemay005 | The screening period/baseline period last about 14 day, and the observation period last about 11 day. The specimen collecting time and observation period may be adjusted appropriately according to the test results.
  peak concentration (Cmax)
pharmacokinetic (PK) profile of Hemay005 | The screening period/baseline period last about 14 day, and the observation period last about 11 day. The specimen collecting time and observation period may be adjusted appropriately according to the test results.
  time-to-peak (Tmax)
pharmacokinetic (PK) profile of Hemay005 | The screening period/baseline period last about 14 day, and the observation period last about 11 day. The specimen collecting time and observation period may be adjusted appropriately according to the test results.
  area under the curve (AUC0-t and AUC0-∞)
pharmacokinetic (PK) profile of Hemay005 | The screening period/baseline period last about 14 day, and the observation period last about 11 day. The specimen collecting time and observation period may be adjusted appropriately according to the test results.
  half-life (t1/2)
pharmacokinetic (PK) profile of Hemay005 | The screening period/baseline period last about 14 day, and the observation period last about 11 day. The specimen collecting time and observation period may be adjusted appropriately according to the test results.
  apparent clearance (CL/F)
pharmacokinetic (PK) profile of Hemay005 | The screening period/baseline period last about 14 day, and the observation period last about 11 day. The specimen collecting time and observation period may be adjusted appropriately according to the test results.
  apparent volume of distribution (Vd/F)
pharmacokinetic (PK) profile of Hemay005 | The screening period/baseline period last about 14 day, and the observation period last about 11 day. The specimen collecting time and observation period may be adjusted appropriately according to the test results.
  mean residence time (MRT0-t)

CONTACTS AND LOCATIONS:
Overall Officials: YanMei Liu, Principal Investigator — Shanghai Xuhui District Central Hospital; GangYi Liu, Principal Investigator — Shanghai Xuhui District Central Hospital
Locations (1):
- Shanghai Xuhui Central Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No